CLINICAL TRIAL: NCT02433119
Title: A Multi-center, Randomized, Double-blind, Phase IV Clinical Trial to Compare the Efficacy and Safety of OROSARTAN® Tablet 5/160mg Versus CODIOVAN® Tablet 160/12.5mg in Patients With Essential Hypertension Uncontrolled With Valsartan 160mg Monotherapy
Brief Title: The Efficacy and Safety of OROSARTAN® Versus CODIOVAN® in Patients With Essential Hypertension Uncontrolled With Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORT_EH_IV
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Amlodipine orotate & Valsartan (Experimental): Amlodipine orotate 6.91mg (5mg as amlodipine) and Valsartan 160 mg, tablet, once a day for 8 weeks
  Interventions: Drug: OROSARTAN® 5/160mg
- Valsartan & Hydrochlorothiazide (Active Comparator): Valsartan 160mg and Hydrochlorothiazide 12.5mg, tablet, once a day for 8 weeks
  Interventions: Drug: CODIOVAN® 160/12.5mg

INTERVENTIONS:
Drug: OROSARTAN® 5/160mg
  Arms: Amlodipine orotate & Valsartan
Drug: CODIOVAN® 160/12.5mg
  Arms: Valsartan & Hydrochlorothiazide

SUMMARY:
A multi-center, randomized, double-blind, phase IV clinical trial to compare the efficacy and safety of OROSARTAN® tablet 5/160mg versus CODIOVAN® tablet 160/12.5mg in patients with essential hypertension uncontrolled with valsartan 160mg monotherapy

ELIGIBILITY:
Inclusion Criteria:

* 19 aged or over
* A patient who was diagnosed with essential hypertension at screening(Visit 1)
* A patient understood objective of this clinical trial and gave their written informed consent voluntarily

Exclusion Criteria:

* A patient with severe hypertension(MSSBP≥200mmHg or MSDBP≥120mmHg) at Visit 1
* A subject with difference(as MSSBP≥20mmHg or MSDBP≥10mmHg) in blood pressure between right and left arm at screening evaluation
* Medical history or evidence of a secondary form of hypertension
* A subject with history of hypersensitivity to CCB(Calcium Channel Blocker), ARB(Angiotensin II Receptor Blocker) or sulfonamide

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Mean Sitting Diastolic Blood Pressure (MSDBP) | Baseline, Week 8

SECONDARY OUTCOMES:
Change from baseline in MSDBP | Baseline, Week 4
Change from baseline in Mean Sitting Systolic Blood Pressure (MSSBP) | Baseline, Week 4 and 8
Control rate in blood pressure | Baseline, Week 8
  Rate of patients who achieved target blood pressure(MSDBP<90mmHg and MSSBP<140mmHg)
Responder rate in blood pressure | Baseline, Week 8
  Rate of patients who achieved MSDBP≥10mmHg and MSSBP≥20mmHg decrease compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Hospital, Incheon, South Korea